CLINICAL TRIAL: NCT02450188
Title: An Integrated Approach With Vardenafil Orodispersible and Cognitive-behavioral Sex Therapy for the Treatment of Erectile Dysfunction (STEDOV)
Brief Title: Vardenafil and Cognitive-behavioral Sex Therapy for the Treatment of Erectile Dysfunction (STEDOV)
Acronym: STEDOV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, Full Professor of Endocrinology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANDRO-AOUC-2014-02
Record Dates: First submitted 2014-12-11; First posted 2015-05-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; PDE5 inhibitors; Cognitive-behavioral Sex Therapy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vardenafil (Active Comparator): The study includes a total period of 10 week with a total of 3 visits for vardenafil Group (at the beginning, at 5th week and at the end). In this study we used Vardenafil 10 mg orodispersible tablets. These are the only orodispersible tablets on commerce indicated for the treatment of ED. Male patients will begin taking Vardenafil 10 mg orodispersible tablets 2 times a week for 10 weeks.
  Interventions: Drug: Vardenafil
- vardenafil+cbst (Active Comparator): The study includes a total period of 10 week with a total of 10 visits for vardenafil+cbst Group (one weekly visit).
  Male patients will begin taking Vardenafil 10 mg orodispersible tablets 2 times a week for 10 weeks.CBST interventions used in this study includes: psycho-educational interventions on ED maintaining, on anxiety's role and sexual homework. This course is structured in 10 weekly meetings.
  Interventions: Drug: Vardenafil; Behavioral: CBST

INTERVENTIONS:
Drug: Vardenafil — In this study we used Vardenafil 10 mg orodispersible tablets. These are the only orodispersible tablets on commerce indicated for the treatment of ED. We choose this kind of tablets because of their easy way of assumption that can also have a minor psychological impact on patients.
  Male patients will begin taking Vardenafil 10 mg orodispersible tablets 2 times a week for 10 weeks.
Behavioral: CBST — The CBST cognitive intervention, in according with Beck (1976), includes to help patients and their partners to gain a commonsense understanding and reframe their problems.
  On the other side, the CBST behaviour intervention, how described by Meichenbaum (1993), is a method to teach patients to practice different behaviours that allows the replacement of the compromised behaviour with a functional one.
  CBST interventions used in this study includes: psycho-educational interventions on ED maintaining, on anxiety's role and sexual homework. This course is structured in 10 weekly meetings. Male patients will begin taking Vardenafil 10 mg orodispersible tablets 2 times a week for 10 weeks.
  Arms: vardenafil+cbst

SUMMARY:
The aim of the present study is to evaluate the efficacy of a combined approach with Vardenafil orodispersible and Cognitive Behavioural Sex Therapy in the treatment of Erectile Dysfunction, compared to medical only treatment, in terms of quality and duration of erection and couple's sexual satisfaction.

DETAILED DESCRIPTION:
This is a randomized controlled study involving 30 subjects with ED, and their partners, seeking medical care for sexual dysfunction at Sexual Medicine and Andrology Unit of Florence's University, Florence, Italy.

Couples were informed that both partners must attend all treatment appointments.

After signed their informed consent form, couples were randomly assigned to two different groups (2:1 ratio), Vardenafil (Group A) or Vardenafil + CBST (Group B), using a computer generated random code.

Couples were randomized for patient's age, partner's age and relationship span, in order to create two homogeneous group.

The study includes a total period of 10 week with a total of 3 visits for Group A (at the beginning, at 5th week and at the end) and with a total of 10 visits for Group B (one weekly visit).

Ethics The ethic committee for clinical trials approved the study protocol, and all patients and their partners provided signed, written, informed consent. The study was conducted in accordance with regulatory standards of Good Clinical Practice and the Declaration of Helsinki (1996).

Participants This study involved 30 male patients with ED, and their partners, both aged > 18 years and in a stable heterosexual relationship (> 6 months), seeking medical care for sexual dysfunction at Andrology Unit of University of Florence, Florence, Italy.

Couples were excluded from participation if man had unstable medical conditions, prior pelvic surgery or trauma, spinal cord injury, prostate surgery or radiation, diabetes mellitus, neurogenic trauma, retinitis pigmentosa, Peyronie's disease, multiple sclerosis, substance abuse disorder, significant mental health problems requiring psychotropic drugs, or were receiving medication for heart disease/angina (especially nitrates) or vascular disease.

Testosterone levels has been considered normal for plasma levels ≥ 12 nmol/L and/or calculated free testosterone≥ 225 pmol/L. When a diagnosis of hypogonadism was made, an adequate testosterone replacement therapy was assessed.

Patients with an artheriogenic ED (assessed with peak systolic velocity at penile colour doppler ultrasound after PGE1 stimulation, considered normal for data ≥ 25 cm/sec ) were excluded.

The investigators also excluded couples including women with primary sexual dysfunction, as dyspareunia, anorgasmia or vaginismus; substance abuse disorder and/or with significant mental health problems requiring psychotropic drugs. The presence of substance abuse or mental health problems was assessed by clinical interviews by a mental health specialist.

Study Procedures Before starting any treatment and before any specific diagnostic procedures, male patients were interviewed by the sexual medicine specialist using SIEDY structured interview. This is a 13-item interview previously validated which identifies and quantifies the contribution of organic, relational and intra-psychic domains of ED.

Patients were also required to provide basic laboratory examinations (including the evaluation of LH, total testosterone, SHBG, glycemia, FSH, TSH, total cholesterol, HDL, PSA, PRL, triglycerides) and to perform a Colour-Doppler Ultrasound (CDU) study of penis.

After completion of this screening by the andrologist, couples were randomly assigned to either Group A for monotherapy with Vardenafil orodispersible or to Group B for the combining treatment with Vardenafil orodispersible and CBST.

The outline of both Group procedures is presented respectively in Table 1 and Table 2.

The CBST cognitive intervention, in according with Beck, includes to help patients and their partners to gain a commonsense understanding and reframe their problems.

On the other side, the CBST behaviour intervention, how described by Meichenbaum, is a method to teach patients to practice different behaviours that allows the replacement of the compromised behaviour with a functional one.

CBST interventions used in this study includes: psycho-educational interventions on ED maintaining, on anxiety's role and sexual homework. This course is structured in 10 weekly meetings.

Materials All participants completed questionnaires at week 1 (before starting treatment), week 5 (in mid of treatment) and week 10 (last session).

Both, male and female, completed the International Index of Erectile Fuction (IIEF-15), the Index of Sexual Satisfaction (ISS) and the Middelsex Hospital Questionnaire (MHQ).

IIEF-15 was used to evaluate male erectile function (erectile function domain, EF) and both male and female sexual satisfaction (intercourse satisfaction, IS domain, and overall satisfaction, OS domain). In fact, even if IIEF-15 has been designed in order to evaluate male sexual function, the investigators also asked the female partner to complete this interview, in order to capture their perception of their partner's erectile function and their own satisfaction.

Couple's sexual satisfaction was also assessed using the ISS, an instrument that assesses any sexual couple's dissatisfaction. The MHQ was used to assess any underlying psychopathology in both partners. Female partners also completed the Female Sexual Function Index (FSFI), to assess their sexual function at the beginning and at the end of treatment. The Authors didn't use the FSFI to exclude sexual female dysfunction because of, in according with previous researches, women who report a partner with ED show significantly lower FSFI scores than women who don't report ED in their partner.

Medicament In this study Vardenafil 10 mg orodispersible tablets were used. These are the only orodispersible tablets on commerce indicated for the treatment of ED. This kind of tablets were chosen because of their easy way of assumption that can also have a minor psychological impact on patients.

Male patients will begin taking Vardenafil 10 mg orodispersible tablets 2 times a week for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* This study involved 30 male patients with ED, and their partners, both aged > 18 years and in a stable heterosexual relationship (> 6 months), seeking medical care for sexual dysfunction at Andrology Unit of University of Florence, Florence, Italy

Exclusion Criteria:

* Couples were excluded from participation if man had unstable medical conditions
* Prior pelvic surgery or trauma
* Spinal cord injury
* Prostate surgery or radiation
* Diabetes mellitus
* Neurogenic trauma
* Retinitis pigmentosa
* Peyronie's disease
* Multiple sclerosis
* Substance abuse disorder
* Significant mental health problems requiring psychotropic drugs, or were receiving medication for heart disease/angina (especially nitrates) or vascular disease.
* Testosterone levels has been considered normal for plasma levels ≥ 12 nmol/L and/or calculated free testosterone≥ 225 pmol/L.
* When a diagnosis of hypogonadism was made, an adequate testosterone replacement therapy was assessed.
* Patients with an artheriogenic ED (assessed with peak systolic velocity at penile colour doppler ultrasound after PGE1 stimulation, considered normal for data ≥ 25 cm/sec ) were excluded.
* We also excluded couples including women with primary sexual dysfunction, as dyspareunia, anorgasmia or vaginismus; substance abuse disorder and/or with significant mental health problems requiring psychotropic drugs.
* The presence of substance abuse or mental health problems was assessed by clinical interviews by a mental health specialist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
erectile function | Time0= at the beginning of treatment, Time 1 = after 5 weeks of treatment and Time 2= after 10 weeks of treatment
  we evaluate change in IIEF-15 erectile function domain from the beginning to the end of treatment (T0 vs.T2)
overall satisfaction | Time0= at the beginning of treatment, Time 1 = after 5 weeks of treatment and Time 2= after 10 weeks of treatment
  we evaluate change in IIEF-15 overall satisfaction domain from the beginning to the end of treatment (T0 vs.T2)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maggi, Principal Investigator — University of Florence
Locations (1):
- Ambulatori Medicina della Sessualità e Andrologia, Florence, Italy

REFERENCES:
- [Background] Dean J, Rubio-Aurioles E, McCabe M, Eardley I, Speakman M, Buvat J, de Tejada IS, Fisher W. Integrating partners into erectile dysfunction treatment: improving the sexual experience for the couple. Int J Clin Pract. 2008 Jan;62(1):127-33. doi: 10.1111/j.1742-1241.2007.01636.x. Epub 2007 Nov 19. PMID 18028387
- [Background] Petrone L, Mannucci E, Corona G, Bartolini M, Forti G, Giommi R, Maggi M. Structured interview on erectile dysfunction (SIEDY): a new, multidimensional instrument for quantification of pathogenetic issues on erectile dysfunction. Int J Impot Res. 2003 Jun;15(3):210-20. doi: 10.1038/sj.ijir.3901006. PMID 12904808
- [Background] Banner LL, Anderson RU. Integrated sildenafil and cognitive-behavior sex therapy for psychogenic erectile dysfunction: a pilot study. J Sex Med. 2007 Jul;4(4 Pt 2):1117-25. doi: 10.1111/j.1743-6109.2007.00535.x. PMID 17627724
- [Background] Montorsi F, Adaikan G, Becher E, Giuliano F, Khoury S, Lue TF, Sharlip I, Althof SE, Andersson KE, Brock G, Broderick G, Burnett A, Buvat J, Dean J, Donatucci C, Eardley I, Fugl-Meyer KS, Goldstein I, Hackett G, Hatzichristou D, Hellstrom W, Incrocci L, Jackson G, Kadioglu A, Levine L, Lewis RW, Maggi M, McCabe M, McMahon CG, Montague D, Montorsi P, Mulhall J, Pfaus J, Porst H, Ralph D, Rosen R, Rowland D, Sadeghi-Nejad H, Shabsigh R, Stief C, Vardi Y, Wallen K, Wasserman M. Summary of the recommendations on sexual dysfunctions in men. J Sex Med. 2010 Nov;7(11):3572-88. doi: 10.1111/j.1743-6109.2010.02062.x. PMID 21040491
- [Result] Boddi V, Castellini G, Casale H, Rastrelli G, Boni L, Corona G, Maggi M. An integrated approach with vardenafil orodispersible tablet and cognitive behavioral sex therapy for treatment of erectile dysfunction: a randomized controlled pilot study. Andrology. 2015 Sep;3(5):909-18. doi: 10.1111/andr.12079. PMID 26311340